CLINICAL TRIAL: NCT06238154
Title: Assessment of Flurbiprofen Tablet and Spray For Postoperative Pain Control In Oral Soft Tissue Wounds: A Randomized Clinical Trial
Brief Title: Flurbiprofen Tablet vs Spray In Oral Soft Tissue Wounds
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, Cennet Neslihan Eroglu, Assoc Prof Dr, Yuzuncu Yil University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 05/25102023
Record Dates: First submitted 2024-01-24; First posted 2024-02-02 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Oral Soft Tissue Conditions; Drug Effect; Drug Use
Keywords: flurpibrofen; oral soft tissue
MeSH Terms: interventions — Flurbiprofen

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: The clinician collecting data from patients was blinded. The researcher who analyzed the results was blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Spray group (Experimental): Spray group consisted of individuals who used flurbiprofen in spray form as a postoperative analgesic
  Interventions: Drug: Flurbiprofen
- Tablet group (Active Comparator): Tablet group consisted of individuals who used flurbiprofen in tablet form as a postoperative analgesic
  Interventions: Drug: Flurbiprofen

INTERVENTIONS:
Drug: Flurbiprofen — The efficacy of two different forms and amounts of active ingredient (100mg tablet vs 25% oral spray) on postoperative pain of different flurbiprofen
  Other Names: Spray flurbiprofen vs Tablet flurbiprofen

SUMMARY:
The amount of active ingredient in tablet form of flurbiprofen is higher than that in the oral spray form. Therefore, based on the hypothesis that the side effects that may occur depending on the dose can be reduced, this clinical study investigated whether tablet and spray form flurbiprofen would have similar effects on postoperative pain in primarily closed soft tissue wounds in the oral region.

DETAILED DESCRIPTION:
In line with the number of patients obtained after sample size calculation, the study was completed on 40 patients who met the inclusion criteria. Patients were healthy, volunteer individuals who required excision of the epulis fissuratum or frenulum with the indication of preprosthetic surgery. 2 groups were formed by simple randomization with 20 patients in the tablet group and 20 patients in the spray group. After the surgical procedure, tablet and spray flurbiprofen were prescribed according to the groups. Apart from these, paracetamol, chlorhexidine gluconate + benzidamine hydrochloride mouthwash were prescribed to all patients as rescue analgesics. The tissue fragments removed from the patients who underwent epulis excision were sent for histopathologic evaluation and confirmed.

ELIGIBILITY:
Inclusion Criteria:

* Provided that those using removable prosthesis had discontinued using the prosthesis 1 month ago (in order to minimize the lesion to be excised), healthy or ASA Class I patients between 40 and 65 years of age, who had the indication of pre-prosthetic surgery due to excision of epulis fissuratum and frenulum

Exclusion Criteria:

* Pregnancy, lactation, and taking contraceptive pills; being allergic to the drug or other NSAIDs to be used in the study; had used steroids or analgesic drugs for any reason for the last 1 month; using psychiatric drugs; those with incomplete data and refused to sign the consent form; those who were extremely afraid and had a gag reflex; those with any gastrointesinal problems; smoking, ASA-2 and ASA-3 patients and those who smoked.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-10-26 (Actual); Primary Completion 2024-01-12 (Actual); Study Completion 2024-01-20 (Actual)

PRIMARY OUTCOMES:
Postoperative pain evaluation with Numeric Rating Scale scores | One week (3, 6, 24, 48, and 72 hours and on the 5th and 7th days)
  The effect of analgesics used in the groups on the level of pain in Numeric Rating Scale (The pain intensity was assessed on a 0-10 ranking scale with 0 representing "no pain" and 10 "most severe pain" ) after soft tissue surgery was investigated.

SECONDARY OUTCOMES:
Rescue analgesic intake | One week
  It was investigated whether rescue analgesics were needed in the groups

OTHER OUTCOMES:
Drug intake amounts | One week
  Assessment of daily analgesic requirement in groups

CONTACTS AND LOCATIONS:
Overall Officials: Cennet N Eroglu, DDS,PhD, Principal Investigator — Yuzuncu Yil University
Locations (1):
- Yuzuncu Yil University, Van, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
After the study is published, the study information will be shared with the researchers who request it, taking into account the right to protect personal data
Supporting Information: Study Protocol, ICF, CSR
Time Frame: IPD and documents will be available for sharing 1 year after publication for a period of 2 years. Access to the IPD and documents will be open on the IPDShare website with registration. The information will be freely available and can be used for any purpose. There will not be any review process or no Data Use Agreement will be necessary.
Access Criteria: IPD and documents will be available for sharing 1 year after publication for a period of 2 years. Access to the IPD and documents will be open on the IPDShare website with registration. The information will be freely available and can be used for any purpose. There will not be any review process or no Data Use Agreement will be necessary.